CLINICAL TRIAL: NCT04928339
Title: Pecto-Intercostal Fascial Plane Block for Enhanced Recovery After Cardiac Surgery
Brief Title: Pecto-Intercostal Fascial Plane Block Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-0111; Protocol Version 01/11/2021 (Other: UW Madison); A530900 (Other: UW Madison); SMPH/ANESTHESIOLOGY (Other: UW Madison)
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Surgery; Opioid Use, Unspecified
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: prospective, single-center, randomized, double-blind, controlled trial
Who Masked: Participant, Care Provider
Masking Description: Each study participant and OR anesthesia team, cardiac surgery team, cardiothoracic ICU team, and nursing staff caring for the participant will be blinded to the study drug the patient received. However, the anesthesia provider performing the block (separate from the provider caring for the patient in the operating room) will not be blinded to the study drug injected and will have access to all monitors deemed appropriate by the primary team caring for the participant.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PIFB intervention (Experimental): bilateral PIFB with a mixture of standard 0.25% bupivacaine (15 mL) and 133 mg liposomal bupivacaine (10mL)
  Interventions: Drug: Bupivacaine Injection; Drug: Liposomal bupivacaine
- Saline Control (Sham Comparator): bilateral PIFB with 25 mL saline only
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Bupivacaine Injection — 10mL of 0.25% bupivacaine
  Arms: PIFB intervention
Drug: Liposomal bupivacaine — 15mL of 133mg liposomal bupivacaine
  Arms: PIFB intervention
Other: Saline — 25mL saline control
  Arms: Saline Control

SUMMARY:
This study is being done to see if bilateral pecto-intercostal fascial plane blocks (PIFB) with a mixture of liposomal and standard bupivacaine decrease pain and opioid requirements in patients undergoing cardiac surgery via median sternotomy compared to controls (sham blocks with saline). 100 participants will be recruited and can expect to be on study for 100 days.

DETAILED DESCRIPTION:
Thousands of heart surgeries are performed every day in the United States. Unattenuated perioperative pain has been shown to contribute to increased morbidity, mortality, length of stay, and healthcare costs. Practice guidelines from the American Society of Regional Anesthesiologists recommend pre-incision techniques to reduce perioperative pain, however in cardiac surgery, there are no commonly used techniques to follow this recommendation. The PIFB is a newly described fascial plane block and existing literature supports the safety and efficacy of the PIFB in cardiac surgery patients. However, there are no randomized controlled trials evaluating this technique with a long-acting depot local anesthetic.

The purpose of this study is to determine whether bilateral pecto-intercostal fascial plane blocks with liposomal bupivacaine decrease pain and opioid requirements in patients undergoing cardiac surgery via median sternotomy compared to controls (sham blocks with saline). The primary hypothesis is that patients receiving effective regional anesthesia with liposomal bupivacaine via PIFB will demonstrate a clinically significant (25%) reduction in total daily opioid consumption through 72 hours postoperatively compared to patients receiving standard of care without effective regional anesthesia (saline only via PIFB).

This study is a prospective, single-center, randomized, double-blind, controlled trial to evaluate whether bilateral pecto-intercostal fascial plane blocks with liposomal and standard bupivacaine decrease pain and opioid requirements in patients undergoing cardiac surgery via median sternotomy compared to controls (sham blocks with saline).

The participants will be randomized to receive bilateral PIFB with a mixture of standard and liposomal bupivacaine or bilateral PIFB with saline only. Recovery characteristics, including opioid consumption, pain scores, duration of mechanical ventilation, ICU length of stay, hospital length of stay, side effects, and chronic opioid use will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Participant provides consent to participate in study
* Ideal body weight (IBW) is >50kg
* Participant is planned to undergo coronary artery bypass graft or single valve repair/replacement surgery via median sternotomy
* Participant is undergoing an elective procedure

Exclusion Criteria:

* Participant is unable or unwilling to give consent
* Non-English speaking
* Known or believed to be pregnant or is currently breastfeeding
* Participant is a prisoner
* Clinically unstable per discretion of the Investigator
* Participant requires urgent/emergent surgery
* History of previous sternotomy
* Preoperative coagulopathy (INR >1.4, platelets <100,000) or ongoing anticoagulation or anti-platelet therapy (except aspirin 81mg)
* Allergy or sensitivity to amide-type local anesthetics, dexmedetomidine or ketamine
* Participant has decompensated heart failure
* Severe left ventricle dysfunction (defined quantitatively as an ejection fraction of less than or equal to 35%) or right ventricle dysfunction (defined qualitatively as "severe")
* Diagnosis of cirrhosis or end-stage liver disease
* Requires the use of mechanical circulatory support pre-operatively
* Participant uses chronic opioids (meaning at the time of the preoperative screening evaluation by the study team, the patient is prescribed and taking any opioid pain medication)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meyer, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simon ER, Mallery A, Silva J, de Biasi A, Osaki S, Krause BM, Meyer P. Superficial parasternal intercostal plane blocks with liposomal bupivacaine did not significantly reduce opioid use after cardiac surgery: a randomized clinical trial. Reg Anesth Pain Med. 2025 Aug 24:rapm-2025-106952. doi: 10.1136/rapm-2025-106952. Online ahead of print. PMID 40850695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at UW Hospitals and Clinics from March 2022 until September 2023
Period: Overall Study
Arm/Group | PIFB Intervention | Saline Control
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PIFB Intervention | Saline Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.50 [57.25 to 70.00] | 64.00 [57.00 to 69.75] | 64 [57.00 to 70.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 36 | 43 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 35 | 33 | 68
  Unknown or Not Reported | 8 | 15 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 33 | 68
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 8 | 15 | 23
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption 72 Hours Post-operatively
Description: Total opioid consumption during the initial 72 hours post-operatively will be measured in morphine milligram equivalents (MME) and compared between groups.
Time Frame: up to 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
morphine milligram equivalents | 165.00 [102.97 to 283.80] | 205.05 [144.94 to 280.80]

2. Secondary Outcome: Total Intraoperative Opioid Consumption
Description: Total intraoperative opioid consumption will be measured in morphine milligram equivalents (MME) and compared between groups.
Time Frame: intraoperative period ranging from anesthesia start time to anesthesia end time
Measure: Median (Full Range); unit: morphine milligram equivalents
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
morphine milligram equivalents | 267.50 [180.75 to 305.40] | 229.80 [176.70 to 284.85]

3. Secondary Outcome: Daily Median Pain Scores First 72 Hours Postoperatively Number of Participants Experiencing Low, Medium or High Pain for up to 72 Hours Post-op
Description: Pain will be assessed, according to standard of care, every 4 hours using the 11-point Numerical Rating Scale (NRS), beginning at time 0 (arrival to ICU). Each patient's pain scores (higher scores indicate worse pain) within each postoperative day will be averaged, and the mean pain scores during each day and throughout the first 72 hours will be compared between the intervention and control groups. Median pain scores at 24, 48 and 72 hours post-op will be interrogated.
  Participants described their pain as low (range of 0-4), medium (range of 5-7) or high (range of 8-10).
Time Frame: data collected immediately post-op, 24 hours, 48 hours, and 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
Participants
  Median Pain at 72 hours post-operatively: low pain | 46 | 47
  Median Pain at 72 hours post-operatively: medium pain | 2 | 1
  Median Pain at 72 hours post-operatively: high pain | 2 | 2
  Median pain scores at 48 hours post-operatively post-op: low pain | 3 | 4
  Median pain scores at 48 hours post-operatively post-op: medium pain | 19 | 22
  Median pain scores at 48 hours post-operatively post-op: high pain | 28 | 24
  Median pain scores at 24 hours post-operatively: low pain | 2 | 2
  Median pain scores at 24 hours post-operatively: medium pain | 17 | 16
  Median pain scores at 24 hours post-operatively: high pain | 31 | 32
  Median Pain immediately post-operatively: low pain | 2 | 0
  Median Pain immediately post-operatively: medium pain | 7 | 7
  Median Pain immediately post-operatively: high pain | 41 | 43

4. Secondary Outcome: Maximum Pain Scores up to 72 Hours Postoperatively
Description: Pain will be assessed, according to standard of care, every 4 hours using the 9-point Numerical Rating Scale (NRS) where higher score indicate worse pain, beginning at time 0 (arrival to ICU). The number of Participants reporting a Maximum pain score at 72 hours postoperatively will be reported. Participants described their pain as low (range of 0-4), medium (range of 5-7) or high (range of 8-9).
Time Frame: up to 72 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
Participants
  High Pain | 29 | 25
  Medium Pain | 19 | 22
  Low Pain | 2 | 3

5. Secondary Outcome: Pain Score at 90 Days Postoperatively
Description: Pain will be assessed, according to standard of care, every 4 hours using the 11-point Numerical Rating Scale (NRS) where higher score indicate worse pain. Pain at 90 days postoperative will be surveyed by phone. Pain will be assessed participants described their pain as low (range of 0-4), medium (range of 5-7) or high (range of 8-10).
Time Frame: up to 90 days post-op
Measure: Median (Inter-Quartile Range); unit: pain score units on a scale
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
pain score units on a scale
  Within 24 hours, worst pain | 3 [1 to 5] | 2 [1 to 3]
  Within 24 hours, least pain | 0 [0 to 2] | 0 [0 to 1]
  Within 24 hours, average pain | 2 [0 to 4] | 1 [0 to 2]

6. Secondary Outcome: Daily Opioid Consumption up to 72 Hours Postoperatively
Description: Daily opioid consumption during the initial 72 hours postoperatively will be measured in milligrams of morphine equivalents and compared between groups.
Time Frame: up to 72 hours post-op
Measure: Median (Inter-Quartile Range); unit: milligrams of morphine equivalents
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
milligrams of morphine equivalents
  Opioid Consumption from 0 to 24 hours post-operatively | 90 [52.80 to 135.60] | 103.80 [73.43 to 137.02]
  Opioid Consumption between 24-48 hours post-operatively | 58.35 [37.50 to 79.95] | 75.00 [29.55 to 105.00]
  Opioid Consumption between 48-72 hours post-operatively | 26.25 [7.88 to 45.00] | 30.00 [0.00 to 60.00]

7. Secondary Outcome: Hours of Mechanical Ventilation After ICU Admission
Description: Duration of mechanical ventilation will be measured by hours of mechanical ventilation after admission to the ICU.
Time Frame: up to 72 hours post-op
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
hours | 4.03 [3.03 to 6.32] | 4.46 [2.98 to 8.11]

8. Secondary Outcome: Number of Postoperative Days Until the First Bowel Movement
Description: Return of bowel function will be measured in the number of postoperative days until the first bowel movement.
Time Frame: up to 72 hours post-op
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
days | 2.81 [2.19 to 3.00] | 2.60 [2.06 to 2.99]

9. Secondary Outcome: Number of Participants Reporting Postoperative Delirium Episodes Per the Confusion Assessment Method for the ICU (CAM-ICU)
Description: Postoperative delirium episodes will be measured according to standard of care by utilizing the CAM-ICU assessment every 8-12 hours. The CAM-ICU determines either 'yes' or 'no' the participant is experiencing delirium. The number of of delirium episodes within 72 hours post-op will be determined.
Time Frame: up to 72 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
Participants | 5 | 8

10. Secondary Outcome: Number of Hours That the Patient is in the ICU
Description: Duration of ICU stay will be measured by the number of hours that the patient is in the ICU until an order is placed for transfer to a lower level of care.
Time Frame: up to 72 hours post-op
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
hours | 20.94 [17.38 to 23.07] | 20.00 [17.28 to 24.32]

11. Secondary Outcome: Number of Post-operative Days Until the Patient is Discharged
Description: Duration of hospital stay will be measured by the number of post-operative days until the patient is discharged.
Time Frame: Up to 7 days
Measure: Median (Full Range); unit: days
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
days | 4.60 [3.84 to 5.68] | 4.51 [3.89 to 5.77]

12. Secondary Outcome: Count of Participants Using Opioids at 90 Days Postoperatively
Description: Patient use of opioids at 90 days will be obtained by phone call.
Time Frame: up to 90 days post-op
Measure: Number; unit: count of participants
Arm/Group | PIFB Intervention | Saline Control
Number analyzed (Participants) | 50 | 50
count of participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Participants were followed for up to 90 days following enrollment.
Arm/Group | PIFB Intervention | Saline Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT04928339/Prot_SAP_ICF_003.pdf